CLINICAL TRIAL: NCT01679925
Title: Qualitative Assessment of the Psychosocial Impact of Early Puberty in Girls Aged 6 to 8 Years
Brief Title: Psychosocial Impact of Early Puberty in Girls Aged 6 to 8 Years
Acronym: PUPSY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P111010
Record Dates: First submitted 2012-07-25; First posted 2012-09-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2012-07

CONDITIONS: Early Puberty
Keywords: Early puberty; Psychosocial impact; Qualitative assessment
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
GnRH agonists are used in the treatment of precocious puberty in order to improve adult height.However,the psychosocial impact of precocious puberty is often used by the clinician at diagnosis to justify treatment, but can not yet be properly assessed. It can not be considered as a rational neither for the indication to treatment, nor to assess its potential efficacy.

The overall objective of this work is to improve the conditions leading to the therapeutic decision and the procedures for monitoring girls with idiopathic central precocious puberty.

DETAILED DESCRIPTION:
During the day hospital, the diagnostic workup for precocious puberty will be performed and include:

* A clinical examination with pubertal stage assessment.
* A GnRH test
* A Pelvic ultrasound
* An MRI will be performed later after the results of GnRH test confirming precocious central puberty.

These reviews are conducted as part of usual care and are required to validate the inclusion criteria of patients.

The CBCL questionnaire will be completed by patient's parents and the first semi-structured interview will be conducted by a sociologist assisted by the psychologist, dedicated to the study.

Patient's follow-up will be planned 6 months after inclusion, including similar investigations (except MRI).

ELIGIBILITY:
Inclusion Criteria:

* 6 to 8 years old girls, with idiopathic central precocious puberty defined as:

  * Onset of clinical signs between 6 and 8 years excluded: breast development (Tanner stage S2 or more), possibly with pubic hair or accelerated growth rate.
  * The GnRH test: LH peak> 5 IU / l during the test.
  * Pelvic ultrasound: uterine length> 34 mm
  * The normality of the hypothalamic-pituitary region assessed by magnetic resonance imaging (MRI).
* Parental Informed and written consent

Exclusion Criteria:

* Parents and / or children do not speak French
* Other chronic disease
* The child does not benefit of the French social security cover

Ages: 6 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be offered to all children and families who visit in a day hospital in the pediatric endocrinology department of Robert Debré Hospital for further assessment of early puberty.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Psychosocial characteristics | 1 day
  * The thematic content related to the perception of early puberty, the factors motivating the consultation, the concerns of families and children, psychosocial characteristics of the subjects received in consultation.
  * The thematic content related to the perception of hormone therapy: identifying the knowledge, concerns and expectations regarding the treatment of precocious puberty.

SECONDARY OUTCOMES:
Child Behavior Checklist | 1 day
  Quantitative data on the psychosocial status of patients will be collected as a self-administered questionnaire: the Child Behavior Checklist (CBCL) that is validated.
Evolution at 6 months | 6 months
  Changing views of qualitative and quantitative data will be followed six months after the diagnosis of precocious puberty, with or without treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique SIMON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Paris, France